CLINICAL TRIAL: NCT01115166
Title: Blood Volume and Fluid Kinetics in Patients Undergoing Extracorporal Circulation
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Joachim Zdolsek, MD, PhD, University Hospital, Linkoeping
Other Study IDs: BVECC
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-09

CONDITIONS: Blood Volume, Extravasation
Keywords: blood volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery: Patients subjected to open cardiac surgery with the help of extracorporal circulation.

SUMMARY:
In patients undergoing extracorporal circulation during cardiac operation, the hemoglobin is subjected to large changes. The purpose of this study is to see if it is possible with the help of volume kinetic techniques to use these variations to measure blood volume and fluid escape from the intravascular volume.

DETAILED DESCRIPTION:
In many clinical situations, such as extensive surgery, it is of value to determine blood volume and rate of fluid loss from the intravascular space, since hypo- and hypervolemia are combined with increased morbidity and mortality. In this study we which to use the large variations in hemoglobin during extracorporal to calculate both these variables.

Hemoglobin is measured every 5 minutes during one hour beginning shortly before start of the heart-lung machine. When the extracorporal circulation begins the hemoglobin decreases due to the quick mix and dilution of the priming fluid from the heart-lung machine with the patients blood.

From the amount of priming fluid and the fall of the hemoglobin, the blood volume can be calculated. If no further fluid is given the next 20 to 30 minutes, the hemoglobin concentration will in most cases increase as a result of the fluid loss from the vascular space. This increase in combination with the diureses can be used to calculate the intravascular fluid loss to the interstitium during surgery.

Sodium concentration will also be measured in parallel with the hemoglobin concentration.

The Sodium concentrations in combination with given and excreted (urine)Sodium can be used in a mass balance to calculate if intracellular edema is induced.

ELIGIBILITY:
Inclusion Criteria:

* open heart surgery, with extracorporal circulation
* consent to participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients subjected to open cardiac surgery, with the help of extracorporal circulation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Zdolsek, MD, PhD, Principal Investigator — University Hospital, Linköping, Sweden
Locations (1):
- University Hospital, Thoracic operation ward, Linköping, Linkoeping, Sweden

REFERENCES:
- [Derived] Tornudd M, Hahn RG, Zdolsek JH. Fluid distribution kinetics during cardiopulmonary bypass. Clinics (Sao Paulo). 2014 Aug;69(8):535-41. doi: 10.6061/clinics/2014(08)06. PMID 25141112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2010 to September 2010 at thoracic surgery department
Pre-assignment Details: Included patients (10). All participated in the study.
Period: Overall Study
Arm/Group | Cardiac Surgery
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Surgery
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 71.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  Sweden | 10

OUTCOME MEASURES:

1. Primary Outcome: Blood Volume
Description: volume kinetic technique: During start of cardio pulmonary by-pass a known amount of fluid will expand the blood volume and dilute the hemoglobin.
  1. The hemoglobin variation is used to calculate the blood volume. The last hemoglobin value before CPB and the hemoglobin value directly after start (extrapolated from the following 30 minutes after start) of CPB are used in the calculation.
  2. The value for the blood volume directly prior to CPB will be influenced by intra venous fluids given during early stages of the anesthesia.
  To achieve the blood volume prior to anesthesia a hemoglobin value before anesthesia and the last hemoglobin value before CPB are used to correct the blood volume calculation. In this way blood volume prior to anaesthesia can be calculated.
Time Frame: 30 minutes after start of CPB
Population: The study was mainly an observational study, and 10 patients was regarded as a sufficient number to register general changes.
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Cardiac Surgery
Number analyzed (Participants) | 10
Litre | 4.61 (0.86)

2. Secondary Outcome: Intracellular Edema
Description: Mass balance based on repeated Sodium concentration, fluid volume given, given and excreted Sodium.
  A positive value indicating intracellular fluid accumulation and a negative value indicating cell dehydration. This is the change that will occur during the first 30 min after start of cardio pulmonary bypass.
Time Frame: 30 minutes after CPB
Population: Mainly observational. 10 patients were regarded to be a sufficient number to se a tendency.
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Cardiac Surgery
Number analyzed (Participants) | 10
Litre | -0.33 (0.557)

3. Other Pre Specified Outcome: Fluid Extravasation
Description: Rate of fluid transfer from the intravascular to the extravascular compartment during two distribution half-times. Graph derived from the hemoglobin change during 20 to 30 minutes after start of cardio pulmonary by-pass.
Time Frame: Two distribution half-times. Approximately 16 minutes.
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: mL/kg/min
Arm/Group | Cardiac Surgery
Number analyzed (Participants) | 10
mL/kg/min | 0.38 (0.24)

ADVERSE EVENTS:
Time Frame: Patients were followed up to 24 hours after CPB. No intervention except additional blood samples was performed, during the CPB.
Arm/Group | Cardiac Surgery
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
The number of patients was small and it was not possible to use a reference method. Standardization was difficult due to the fact that it was a clinical study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No